CLINICAL TRIAL: NCT01254084
Title: Gynostemma Pentaphyllum Tea Improves Insulin Sensitivity in Type 2 Diabetic Patients
Brief Title: Effect of Gynostemma Pentaphyllum Tea in Insulin Sensitivity in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: Karolinska Institutet (Other); Swedish International Development Cooperation Agency (SIDA) (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Diabetes II-Study3; Study 3
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-02

CONDITIONS: Type 2 Diabetes
Keywords: Herbal medicine; Type 2 diabetes; Gynostemma pentaphyllum Tea; Insulin sensitivity;
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo tea (Placebo Comparator): Dietary Supplement: Placebo tea 3 gram twice daily, orally
  Interventions: Dietary Supplement: Placebo tea
- Gynostemma pentaphyllum Tea (Active Comparator): Gynostemma Pentaphyllum tea 3 grams twice daily, orally
  Interventions: Dietary Supplement: Gynostemma Pentaphyllum tea

INTERVENTIONS:
Dietary Supplement: Gynostemma Pentaphyllum tea — 6g/day per oral, twice a day in 10 weeks, 30 minutes before breakfast and dinner
  Other Names: Gynostemma Pentaphyllum extract
  Arms: Gynostemma pentaphyllum Tea
Dietary Supplement: Placebo tea — 6g/day per oral, twice a day in 10 weeks, 30 minutes before breakfast and dinner
  Other Names: Placebo extract
  Arms: Placebo tea

SUMMARY:
The aim of the present study was to investigate the effects of Gynostemma Pentaphyllum tea on insulin sensitivity in drug-naïve type 2 diabetic patients.

DETAILED DESCRIPTION:
In Vietnam, traditional herbal medicines have played a major role in the management of diabetes for centuries. Gynostemma Pentaphyllum (GP) Makino (Family Cucurbitaceae) is a perennial creeping herb growing wild in the mountainous regions of Vietnam, China and some other Asian countries and was widely used in Southeast Asian countries as an herbal medicine and being beneficial for the prevention and treatment of diabetes. We have previously published the evidences that GP tea possessed anti-diabetic effect with good safety data in newly diagnosed T2D patients, and had effect on insulin sensitivity. In addition extract of GP had been shown to reduce both hyperglycemia and hyperlipidemia in diabetic Zucker Fatty rats. So the present study was to investigate the effects of Gynostemma Pentaphyllum tea in insulin sensitivity in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, drug-naive patients with type 2 diabetes
* Fasting plasma glucose: 7-11 mmol/l
* HbA1C: 7-9%.

Exclusion Criteria:

* Type 1 diabetes
* Liver and kidney failure

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Fating plasma glucose, Steady state plasma glucose in Somatostatin-Insulin-Glucose Infusion Test | 10 weeks
  All subjects participated in Somatostatin-Insulin-Glucose Infusion Test (SIGIT), lasting 150 minutes, performed at 8am after an 8-10h overnight fast with only tap water allowed ad libitum. Somatostatin was used to suppress endogenous insulin release, thereby allowing estimation of sensitivity to exogenously administered insulin by measuring blood glucose value at 90, 120 and 150 minute of the test (SIGIT mean).

SECONDARY OUTCOMES:
Liver enzymes (ALT, AST) | 10 weeks
Kidney function (S-creatinine, S-BUN) | 10 weeks
Plasma lipids (TG, Cholesterol, HDL-, LDL-) | 10 weeks
Blood pressure | 10 weeks
Body weight (BMI, hip-waist ratio) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claes-Goran Ostenson, MD, Ph.D, Study Director — Karolinska Institutet
Locations (2):
- Vietnam (2):
  - National Institute of Gerontology, HMU, Hanoi
  - National Institute of Gerontology, Hanoi

REFERENCES:
- [Background] Huyen VT, Phan DV, Thang P, Hoa NK, Ostenson CG. Antidiabetic effect of Gynostemma pentaphyllum tea in randomly assigned type 2 diabetic patients. Horm Metab Res. 2010 May;42(5):353-7. doi: 10.1055/s-0030-1248298. Epub 2010 Mar 8. PMID 20213586
- [Background] Hoa NK, Norberg A, Sillard R, Van Phan D, Thuan ND, Dzung DT, Jornvall H, Ostenson CG. The possible mechanisms by which phanoside stimulates insulin secretion from rat islets. J Endocrinol. 2007 Feb;192(2):389-94. doi: 10.1677/joe.1.06948. PMID 17283239
- [Background] Hoa NK, Phan DV, Thuan ND, Ostenson CG. Screening of the hypoglycemic effect of eight Vietnamese herbal drugs. Methods Find Exp Clin Pharmacol. 2009 Apr;31(3):165-9. doi: 10.1358/mf.2009.31.3.1362514. PMID 19536359
- [Background] Norberg A, Hoa NK, Liepinsh E, Van Phan D, Thuan ND, Jornvall H, Sillard R, Ostenson CG. A novel insulin-releasing substance, phanoside, from the plant Gynostemma pentaphyllum. J Biol Chem. 2004 Oct 1;279(40):41361-7. doi: 10.1074/jbc.M403435200. Epub 2004 Jun 25. PMID 15220351